CLINICAL TRIAL: NCT03054896
Title: Venetoclax Plus Dose-adjusted R-EPOCH or R-CHOP for Richter's Syndrome
Brief Title: A Phase II Study of Venetoclax in Combination With Dose-adjusted EPOCH-R or R-CHOP for Patients With Richter's Syndrome
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Matthew S. Davids, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-596
Record Dates: First submitted 2017-02-10; First posted 2017-02-16 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Richter Syndrome
Keywords: Richter Syndrome
MeSH Terms: interventions — venetoclax; R-CHOP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VR-EPOCH (Experimental): * Standard chemotherapy regimen, DA-EPOCH-R, with a novel oral Bcl-2 inhibitor, venetoclax will be administered to patients
  * Chemotherapy cycles will be administered approximately every 3 weeks
  * Initial venetoclax dose ramp-up will be done in a condensed fashion over approximately 5 days, followed by continuous daily dosing
  Interventions: Drug: Venetoclax; Other: DA-EPOCH-R
- VR-CHOP (Experimental): * Standard chemotherapy regimen, R-CHOP, with a novel oral Bcl-2 inhibitor, venetoclax will be administered to patients
  * Chemotherapy cycles will be administered approximately every 3 weeks
  * Initial venetoclax dose ramp-up will be done in a condensed fashion over approximately 5 days, followed by continuous daily dosing
  Interventions: Drug: Venetoclax; Other: R-CHOP

INTERVENTIONS:
Drug: Venetoclax — Venetoclax is an Antineoplastic Agent; BCL-2 Inhibitor
  Other Names: Venclexta
Other: DA-EPOCH-R — Intensive chemotherapy regiment
  Arms: VR-EPOCH
Other: R-CHOP — Intensive chemotherapy regiment
  Arms: VR-CHOP

SUMMARY:
This research study is evaluating the combination of a study drug, venetoclax, and a standard chemotherapy regimen, R-EPOCH or R-CHOP, as a possible treatment for Richter's Syndrome.

The drugs involved in this study are:

* Venetoclax
* R-EPOCH:

  * Rituximab
  * Etoposide
  * Prednisone
  * Vincristine Sulfate (Oncovin)
  * Cyclophosphamide
  * Doxorubicin Hydrochloride (Hydroxydaunomycin)
* R-CHOP:

  * Rituximab
  * Cyclophosphamide Vincristine
  * Doxorubicin Hydrochloride (Hydroxydaunomycin)
  * Sulfate (Oncovin)
  * Prednisone

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

Tumor cells from patients with Richter's Syndrome are often resistant to chemotherapy. One reason for this may be that a protein called BCL-2 can prevent cancer cells from dying after being exposed to chemotherapy. Venetoclax is an oral drug that specifically targets BCL-2. It has already been shown to be highly effective at killing tumor cells from CLL patients whose cells are resistant to chemotherapy, leading to its FDA (the U.S. Food and Drug Administration) approval for these patients. A small number of patients with Richter's Syndrome have been treated with venetoclax as a single drug, and some of these patients had improvement of their cancer with this treatment.

In this research study, the investigators are looking to see whether adding venetoclax to a standard chemotherapy regimen, R-EPOCH or R-CHOP, will help this chemotherapy work better to more effectively kill tumor cells in patients with Richter's Syndrome. Venetoclax is not approved for Richter's Syndrome or for use in combination with chemotherapy, which is why its use in this trial is considered to be investigational.

ELIGIBILITY:
Inclusion Criteria:

* Must have a confirmed diagnosis of chronic lymphocytic leukemia or small lymphocytic lymphoma as per IW-CLL 2008 criteria (Hallek et al, 2008) with biopsy proven transformation to diffuse large B cell lymphoma (DLBCL), consistent with Richter's Syndrome.
* Age greater than or equal to 18 years. Because CLL and Richter's Syndrome are extremely rare in persons <18 years of age, children are excluded from this study.
* ECOG performance status <2 (see Appendix A)
* Patients must meet the following hematologic criteria at screening, unless they have significant bone marrow involvement of their malignancy confirmed on biopsy:

  * Absolute neutrophil count ≥1000 cells/mm3 (0.5 x 109/L). Growth factor allowed to achieve
  * Platelet count ≥40,000 cells/mm3 (40 x 109/L) independent of transfusion within 7 days of screening
* Subject must have adequate coagulation, renal, and hepatic function, per laboratory reference range at Screening as follows:

  * Creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min using 24-hour urine collection for creatinine clearance
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 × ULN;
  * Bilirubin ≤ 1.5 × ULN;
  * Subjects with Gilbert's Syndrome or resolving autoimmune hemolytic anemia may have a bilirubin up to 3.0 × ULN and are still eligible
* The effects of venetoclax on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Contraception must continue for an additional 30 days post last dose of venetoclax for women, and an additional 90 days post last dose in men. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately and venetoclax must be discontinued immediately.

  * For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception and agreement to refrain from donating eggs, as defined below:
  * Women must remain abstinent or use contraceptive methods with a failure rate of <1% per year during the treatment period and for at least 30 days after the last dose of venetoclax and 12 months after the last dose of chemotherapy, whichever is later. Women must refrain from donating eggs during this same period.
  * A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis). The definition of childbearing potential may be adapted for alignment with local guidelines or regulations. Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
  * For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating sperm, as defined below:
  * With a female partner of childbearing potential who is not pregnant, men who are not surgically sterile must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of <1% per year during the treatment period and for at least 90 days after the last dose of venetoclax or 12 months after completion of chemotherapy, whichever is later. Men must refrain from donating sperm during this same period. With a pregnant female partner, men must remain abstinent or use a condom during the treatment period and for at least 90 days after the last dose of venetoclax or 12 months after the last dose of chemotherapy, whichever is later, to avoid exposing the embryo.
* Patients who have undergone prior allogeneic transplantation are eligible provided they do not have significant active graft versus host disease and that their transplant day 0 is > 6 months from their first dose of chemotherapy
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with the Hodgkin variant transformation of CLL will be excluded
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy or to the chemotherapy drugs used in this study (see Appendix D), unless the antibody can be given through a desensitization program in consultation with an allergist
* Subject has received any of the following within 14 days or 5 drug half-lives (whichever is shortest) prior to the first dose of chemotherapy, or has not recovered to less than Grade 2 clinically significant adverse effect(s)/toxicity(s) of the previous therapy:

  --Any anti-cancer therapy including chemotherapy, biologic agents for anti-neoplastic treatment (e.g. monoclonal antibodies) or radiotherapy, investigational therapy, including targeted small molecule agents. Patients who are currently receiving treatment with ibrutinib or acalabrutinib may continue this agent until the day prior to starting venetoclax, to reduce the risk of tumor flare on treatment cessation.
* Received previous treatment with R-CHOP, R-EPOCH, or R-hyper-CVAD
* History of other malignancies, except:

  * Malignancy treated with curative intent and with no known active disease present before the first dose of study drug and felt to be at low risk for recurrence by treating physician.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated carcinoma in situ without evidence of disease
  * Low-risk prostate cancer on active surveillance
* Concurrent systemic immunosuppressant therapy (eg, cyclosporine A, tacrolimus, etc.) within 28 days of the first dose of study drug.
* Corticosteroids are allowed, but must be dosed at prednisone 20 mg (or equivalent) or lower prior to the start of chemotherapy.
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug.
* Known bleeding disorders (eg, von Willebrand's disease) or hemophilia.
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
* History of human immunodeficiency virus (HIV) or Human T-Cell Leukemia Virus 1 (HTLV-1), or active hepatitis C virus (HCV) or hepatitis B virus (HBV). Patients who are positive for hepatitis B core antibody or hepatitis B surface antigen must have a negative polymerase chain reaction (PCR) result before enrollment, i.e. HBV DNA must be undetectable, provided that they are willing to undergo monthly DNA testing. Those who are PCR positive will be excluded. Patients who are positive for HCV antibody are eligible only if PCR is negative for HCV RNA.
* Any uncontrolled active systemic infection.
* Major surgery within 4 weeks of first dose of study drug.
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 2 or higher congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization.
* Unable to swallow capsules or malabsorption syndrome, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction at time of screening.
* Breastfeeding or pregnant. Serum pregnancy test will be conducted.
* Male subject who is considering fathering a child or donating sperm during the study or for approximately 90 days after the last dose of study drugs.
* Unwilling or unable to participate in all required study evaluations and procedures. Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations)
* Patients receiving any other study agents
* Patients with known CNS involvement
* Baseline QTcF >480 ms. NOTE: This criterion does not apply to patients with a left bundle branch block.
* Patients who require warfarin or other vitamin K antagonists for anticoagulation (other anticoagulants are allowed).
* Concurrent administration of medications or foods that are strong inhibitors or inducers of CYP3A (see Appendix B).
* Patients with ongoing use of prophylactic antibiotics are eligible as long as there is no evidence of active infection and the antibiotic is not a prohibited medication
* Unable to receive prophylactic treatment for pneumocystis, herpes simplex virus (HSV), and herpes zoster (VZV) at start of treatment
* Significant co-morbid condition or disease which in the judgment of the Principal Investigator would place the patient at undue risk or interfere with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Complete Response by 2008 IW-CLL Response Criteria | 2 years
  Complete Response Rate

SECONDARY OUTCOMES:
Partial Response Rate by 2008 IW-CLL Response Criteria | 2 years
  Partial Response Rate
Progression Free Survival | 2 years
  PFS
Overall Survival Rate | 2 years
  OS
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 years
  Treatment-related AEs

CONTACTS AND LOCATIONS:
Overall Officials: Matthew S. Davids, MD, MMSc, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Ohio State University, Columbus, Ohio
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davids MS, Rogers KA, Tyekucheva S, Wang Z, Pazienza S, Renner SK, Montegaard J, Ihuoma U, Lehmberg TZ, Parry EM, Wu CJ, Jacobson CA, Fisher DC, Thompson PA, Brown JR. Venetoclax plus dose-adjusted R-EPOCH for Richter syndrome. Blood. 2022 Feb 3;139(5):686-689. doi: 10.1182/blood.2021011386. PMID 34788401